CLINICAL TRIAL: NCT02537600
Title: Evaluation of Cobimetinib + Vemurafenib Combination Treatment in Patients With Brain Metastasis BRAFV600 Mutated Cutaneous Melanoma
Brief Title: Vemurafenib and Cobimetinib Combination in BRAF Mutated Melanoma With Brain Metastasis
Acronym: CONVERCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-TL-MEL-Th; 2014-001671-30 (EudraCT Number)
Record Dates: First submitted 2015-08-18; First posted 2015-09-01 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2019-01

CONDITIONS: Malignant Melanoma
Keywords: BRAF mutation; Brain metastasis; Cobimetinib + Vemurafenib combination treatment
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cobimetinib + Vemurafenib combination (Experimental): Every patients will be treated with :
  Vemurafenib 1920 mg / day from day 1 to day 28 continuously Cobimetinib 60 mg / day from day 1 to day 21 One cycle = 28 days Intervention = Cobimetinib + Vemurafenib combination treatment. Only one arm.
  Interventions: Drug: Cobimetinib + Vemurafenib combination treatment

INTERVENTIONS:
Drug: Cobimetinib + Vemurafenib combination treatment — Patients will be treated from day 1 to day 28 with Vemurafenib and from day 1 to day 21 with Cobimetinib. Day 1 to Day 28 corresponds to one cycle of treatment.
  Other Names: Vemurafenib = Zelboraf (commercial name); Cobimetinib = code number RO5514041/F04

SUMMARY:
The purpose of this study is to determine wether cobimetinib + vemurafenib combination treatment is effective in the treatment of BRAFV600-mutated melanoma patients with brain metastasis

DETAILED DESCRIPTION:
Patients will be enrolled into 3 cohorts:

* Cohort A : Neurologically asymptomatic patients who have not received prior local treatment ;
* Cohort B. Neurologically asymptomatic patients who have received prior local treatment;
* Cohort C. Neurologically symptomatic patients who have or have not received prior local treatment Every patients will be treated with Vemurafenib 960 mg PO, twice daily from D1 to D28, continuously

Cobimetinib 60 mg PO, once daily, from D1 to D21 - 1 cycle = 28 days

Treatment will be administered until progression (intracranial or extracranial), unacceptable toxicity, withdrawal of consent, death or decision of the treating investigator.

Patients who develop intracranial or extracranial progression and who, in the opinion of the treating investigator, could benefit from continuing treatment may continue treatment with vemurafenib and cobimetinib after approval from the principal investigator.

Patients who discontinue the study treatment will undergo an end-of-treatment visit 30 days after the last dose of vemurafenib and/or cobimetinib.

Patients who discontinue the study treatment for any reason other than progression (e.g. toxicity) must be followed up every 8 weeks unless they withdraw their consent.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Histologically confirmed metastatic cutaneous melanoma, mucous melanoma, or melanoma of unknown primary origin (stage IV).
3. Documented BRAFV600 mutation determined in a hospital center specializing in the molecular genetics of cancer that is certified by the French national cancer institute (INCa).
4. Presence of Brain Metastases (BM) for which surgical resection is not a reasonable treatment option but that may be amenable to treatment with targeted therapy, to be decided in the onco-dermatology and/or neuro-oncology multidisciplinary team meeting (MDTM).
5. At least one measurable BM in at least one dimension between 5 and 40 mm on magnetic resonance imaging (MRI) with gadolinium (modified RECIST 1.1).
6. Patients having previously received a maximum of two systemic therapies during the metastatic phase, except BRAF, Map ERK Kinase (MEK) or Extracellular signal Regulated Kinase (ERK) inhibitors or tyrosine kinase pan-inhibitors (TKIs); prior ipilimumab therapy is allowed if patients have documented cerebral progression 12 weeks after the last injection of treatment and if MRI confirms progression at least 4 weeks later. A period of at least 6 weeks must be observed between the last dose of ipilimumab and the first administration of the study treatments. Prior treatment with anti-programmed cell death (PD)-1 or anti-PD ligand 1 (PD-L1) is allowed.
7. For patients who have received prior whole brain radiotherapy or radiosurgery and/or surgery for BM (cohorts B and C) demonstration of a significant progression of at least one lesion according to RECIST 1.1 criteria, . after at least 4 weeks have elapsed since this treatment has ended, and MRI at inclusion must demonstrate a significant progression of at least one lesion according to RECIST 1.1 criteria.
8. Patients with symptomatic or asymptomatic BM.
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
10. Patients must have recovered from all the side effects (grade ≤ 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events, NCI-Common Toxicity Criteria for Adverse Event (CTCAE), version 4.03) of their most recent systemic or local treatment (except alopecia).
11. Signed and dated informed consent before carrying out any procedures that are specific to the trial and are not procedures (examinations) conducted as part of normal patient care.
12. Patients willing and able to comply with scheduled visits, treatment schedule, laboratory testing and other trial procedures.
13. Negative serum pregnancy test within 10 days of the first dose of the study treatment for women of childbearing age. Women of non-childbearing potential may be included if they are surgically sterile or postmenopausal for ≥ 1 year.
14. Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after the last administration of the study treatment. Effective methods of contraception are defined as those that have a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as injectable implants combined with oral contraception or intra-uterine devices, or as total abstinence in cases where the lifestyle of the patient ensures compliance.
15. Adequate hematologic, renal and hepatic function within 14 days of the administration of treatment:

Hematologic Leucocytes > 2.0 x 109/L Neutrophils > 1.0 x 109/L Hemoglobin (transfusion allowed) > 9 g/dL Platelets > 100 x 109/L Liver Total bilirubin < 1.5 x upper limit of normal (ULN) (< 3.0 mg/dL for patients with Gilbert syndrome) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN if there is liver metastasis) Alkaline phosphatase (ALP) < 3 x ULN (< 5 x ULN if there is liver or bone metastasis) Kidney Creatinine Or creatinine clearance < 1.5 x ULN ≥ 40 mL/min (Cockcroft-Gault formula)

Exclusion Criteria:

1. Uveal melanoma. Patients with mucous melanoma or melanoma of unknown primary origin are eligible if BRAFV600 mutation is confirmed.
2. Symptomatic or diffuse leptomeningeal involvement.
3. Symptoms of uncontrolled intracranial pressure. Increasing corticosteroid dose during the 7 days prior to the first dose of the study treatment is an exclusion criterion. Patients receiving corticosteroids and patients presenting intermittent seizures may be enrolled if the dose of corticosteroids and anti-epileptic treatments has been stable for at least 2 weeks before inclusion.
4. Indication for urgent neurosurgery or radiotherapy.
5. Prior malignancy active within the previous 3 years except for locally curable cancers that have been treated to complete remission or untreated stage I chronic lymphoid leukemia.
6. Known human immunodeficiency virus (HIV) infection.
7. Prior treatment with BRAF, MEK, or ERK inhibitors or pan-TKIs.
8. Concurrent administration of any anticancer therapies other than those administered in this study.
9. Treatment with any cytotoxic and/or investigational drug or targeted therapy within 4 weeks of the first dose of the study treatment, or ipilimumab, anti-PD-1 or anti-PD-L1 immunotherapy within 8 weeks of the study treatment and/or radiation therapy within 2 weeks of the study treatment.
10. Pregnant or breastfeeding women.
11. Refractory nausea and vomiting, intestinal malabsorption, or significant bowel resection that would preclude adequate absorption or cause an inability to swallow tablets.
12. Ulcerative colitis, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticula or other gastrointestinal condition increasing the risk of perforation.
13. Any of the following within the 6 months prior to the first dose of study treatment:

    * myocardial infarction,
    * severe/unstable angina,
    * symptomatic congestive heart failure (New York Heart Association grade ≥2),
    * cerebrovascular accident or transient ischemic attack,
    * pulmonary embolism,
    * grade > 2 hypertension not controlled by medications.
14. History or presence of clinically significant ventricular or atrial arrhythmia ≥ grade 2 (NCI-CTCAE Version 4.03).
15. Corrected QT (cQT) interval ≥ 450 ms and left ventricular ejection fraction (LVEF) below the lower limit of normal (LLN) or < 50% (scintigraphy or ultrasound).
16. History, risk factor or retinal pathology that increases the risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR): evidence of retinal pathology that is considered a risk factor for RVO or CSR, or a history of retinal detachment, central serous chorioretinopathy or retinal vein thrombosis. The risk factors for RVO are listed below:

    * Uncontrolled glaucoma with intraocular pressures > 21 mm Hg,
    * Serum cholesterol ≥ Grade 2 (≥ 7.75 mmol/L),
    * Hypertriglyceridemia ≥ Grade 2 (≥ 3.42 mmol/L),
    * Hyperglycemia (fasting) ≥ Grade 2 (≥ 8.9 mmol/L).
17. Serious or uncontrolled medical disorders that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the patient to follow the protocol, or interfere with the interpretation of study results.
18. Patients Under guardianship or curators, maintenance of justice, non-informed about diagnosis, unable to follow study medical requirement for geographical, social or psychic reasons.
19. Patients with abnormal blood electrolyte test (Ca, Mg, K and Na) that could not be corrected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Complete or partial intracranial response rate in cohort A on the evaluation of each patient's best tumor response by the centralized review committee according to modified Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria. | From baseline up to 36 months

SECONDARY OUTCOMES:
Complete or partial intracranial response rates in cohorts B and C based on the evaluation of each patient's best tumor response by the centralized review committee according to modified RECIST 1.1 criteria. | Up to 36 months
Intracranial duration of response (DR) in cohorts A, B and C. | Up to 36 months
Overall response rate of cohorts A, B and C | Up to 36 months
Overall survival in cohorts A, B and C | Up to 36 months
Frequency of Adverse events | Up to 36 months
Overall duration of response (DR) in cohorts A, B and C. | Up to 36 months
Patient free survival in cohorts A, B and C | Up to 36 months

OTHER OUTCOMES:
Ratio between cerebrospinal fluid concentration and plasmatic exposure of vemurafenib and cobimetinib | At Day15 Cycle 1
BRAF mutation rate in circulating DNA tumor | From baseline up to treatment stop or progression. An average of 8 cycles of treatment is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lesimple, MD, Principal Investigator — Centre Eugène Marquis
Locations (17):
- France (17):
  - CHU de Bordeaux, Bordeaux
  - CHU Ambroise Paré, Boulogne
  - CHU Brest - Hôpital Morvan, Brest
  - CHU Caen - Hôpital Clémenceau, Caen
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU Albert Michallon, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - CHRU Lille, Lille
  - Centre Hospitalier Lyon Sud, Lyon
  - CHU de Nantes, Nantes
  - Groupe Hospitalier l'Archet, Nice
  - Hôîtal St louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Bichat, Paris
  - Centre Eugène Marquis, Rennes
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No